CLINICAL TRIAL: NCT05538624
Title: A Phase 1/2 Open-Label, Multicenter, Dose Escalation and Expansion Study of AVB-001, an Intraperitoneally Administered, Cell-Generated, Human IL-2 Immunotherapy in Patients With Platinum-Resistant, High-Grade, Serous Adenocarcinoma of the Ovary, Primary Peritoneum, or Fallopian Tube
Brief Title: A Study of Intraperitoneally Administered AVB-001 in Patients With Serous Adenocarcinoma of the Ovary
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision to close study
Sponsor: Avenge Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVB-1A-101
Record Dates: First submitted 2022-08-22; First posted 2022-09-14 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Neoplasm, Ovarian; Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Adenocarcinoma Ovary; Serous Adenocarcinoma of Ovary; Serous Adenocarcinoma of Primary Peritoneum; Primary Peritoneal Carcinoma; High Grade Serous Adenocarcinoma
Keywords: Ovarian Cancer; Primary Peritoneum Cancer; Fallopian Tube Cancer; Immunotherapy; IL-2 Immunotherapy; Metastatic Cancer; Human Interleukin 2; Interleukin 2; IL-2; Encapsulated Cell Therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: In this two-part study, Part 1 is the Dose Escalation Phase; Part 2 is the Dose Expansion Phase.
Masking Description: Not applicable in this open-label trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1 escalating AVB-001 between 0.6 and 3.6 ug hIL-2/kg/day; and Part 2 AVB-001 at the MTD/RP2D (Experimental): Part 1: one of four ascending doses of AVB-001 planned for IP, single dose administration at each dose level cohort of the Dose Escalation Phase.
  Part 2: a single dose of AVB-001 at the MTD/RP2D level (determined in Part 1) to be further evaluated in the Dose Expansion Phase.
  Interventions: Drug: AVB-001 (Dose Escalation Phase); Drug: AVB-001 (Dose Expansion Phase)

INTERVENTIONS:
Drug: AVB-001 (Dose Escalation Phase) — One of four ascending doses of AVB-001 planned for IP, single dose administration in each dose level cohort of the Dose Escalation Phase (Part 1).
Drug: AVB-001 (Dose Expansion Phase) — The MTD/RP2D as determined in the Dose Escalation Phase will be further evaluated in the Dose Expansion Phase.

SUMMARY:
This is an open-label, First-in-Human, Phase 1/2, multicenter study to evaluate the safety and efficacy of a single dose of AVB-001. AVB-001 is an encapsulated cell product engineered to produce native human interleukin-2 (hIL-2). It is delivered intraperitoneally (IP) to patients with high grade serous adenocarcinoma of the ovary, primary peritoneum, or fallopian tube.

DETAILED DESCRIPTION:
This is an open-label, First-in-Human, Phase 1/2, multicenter study to evaluate the safety and efficacy of a single dose of AVB-001. AVB-001 is an encapsulated cell product engineered to produce native human interleukin-2 (IL-2). It is delivered intraperitoneally (IP) to patients with high grade serous adenocarcinoma of the ovary, primary peritoneum, or fallopian tube.

The study will be conducted in two parts. Part 1 is the Dose Escalation Phase using a Bayesian optimal interval (BOIN) model-assisted design in which a single dose of 1 of 4 dose levels of AVB-001 will be administered intraperitoneally (IP) in up to 24 patients. The four ascending dose levels of AVB-001 are targeted to produce hIL-2 levels of 0.6, 1.2, 2.4, and 3.6 μg hIL-2/kg/day. The purpose of Part 1 is to determine the maximally tolerated dose (MTD)/recommended Phase 2 dose (RP2D) level.

Part 2 is the Dose Expansion Phase 2 in which a single dose of AVB-001 at the RP2D will be administered in up to 20 additional adult patients with platinum-resistant, high-grade, serous adenocarcinoma of the ovary, primary peritoneum, or fallopian tube. Additional expansion cohorts may be opened in Part 2 either as monotherapy or as an exploratory combination strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed, metastatic or unresectable, platinum-resistant, high-grade, serous adenocarcinoma of the ovary, primary peritoneum, or fallopian tube;

   Note: For the purposes of this study, platinum-resistant is defined as a patient who has received platinum-containing chemotherapy and either has platinum-refractory disease (progressed during initial platinum-based chemotherapy) or resistant disease (relapsed within 6 months of initial platinum-containing chemotherapy) or, if previously with platinum-sensitive disease, has received at least 2 lines of platinum-containing chemotherapy and progressed.

   Note: A pathology report confirming histology will be required for enrollment.
2. Have not received more than 5 lines of prior therapy;
3. May have received poly adenosine diphosphate-ribose polymerase (PARP) inhibitors, bevacizumab (or any other antiangiogenic agent), immunotherapy, or cell therapies. (Patients with germline or somatic breast cancer gene (BRCA) mutations must have progressed or been intolerant to PARP inhibitor therapy);
4. Have an Eastern Cooperative Oncology Group performance status 0 to 1 at Screening;
5. Meet the following laboratory criteria:

   * Absolute neutrophil count >1500/μl;
   * Hemoglobin level ≥9.0 g/dL (transfusion allowed);
   * Platelet count ≥100,000/μl;
   * Creatinine clearance ≥50 mL/minute, measured using the Cockcroft-Gault formula, and serum creatinine ≤1.5 upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) ≤2.5× ULN, aspartate aminotransferase (AST) ≤2.5×ULN; and total bilirubin ≤1.5×ULN (or ≤3×ULN in cases of Gilbert's syndrome); and
   * International normalized ratio <1.5 and activated partial thromboplastin time (or partial thromboplastin time) within normal limits per the institution.

   Note: Patients on direct-acting anticoagulants or other anticoagulation medications are eligible as long as they are able to hold the drug for the laparoscopic procedure on Day 1 per institutional guidance.
6. Have evidence of measurable disease on computed tomography (CT) or magnetic resonance imaging (MRI) scan as defined by RECIST v1.1;

   Note: Measurable disease cannot include a lesion that was biopsied. Patients must, at a minimum, have 1 measurable lesion.

   Note: Patients with IP disease who also have disease involving the pleural cavity or distant metastases will be eligible if they have measurable or evaluable disease in the IP cavity.
7. Are willing and able to provide written informed consent or have a legally authorized representative willing and able to provide informed consent at Screening.

Exclusion Criteria:

1. Have low-grade serous, mucinous, clear cell, or endometrioid adenocarcinoma of the ovary, primary peritoneum, or fallopian tube; carcinosarcoma; or a mixed histology tumor;
2. Have another malignancy or have had a prior malignancy within 3 years prior to the first dose of study drug or any evidence of residual disease from a previously diagnosed malignancy, excluding adequately managed with curative-intent treatment for basal cell carcinoma, squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, cervical carcinoma in situ, melanoma in situ, or ductal carcinoma in situ of the breast;
3. Have a known or suspected allergy to AVB-001 or known or suspected allergy to any components of AVB-001, including alginate or seaweed;
4. Have any condition that, in the opinion of the Investigator, would lead to the inability of the patient to comply with the Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) of IP administered AVB-001 to determine the MTD and RP2D in the Dose Escalation Phase (Part 1) | 4 weeks
Incidence of treatment-emergent adverse events (AEs) and serious AEs (SAEs) of IP administered AVB-001 in the Dose Escalation Phase (Part 1) | 1 year
Investigator-assessed objective response rate (ORR) per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 of IP administered AVB-001 in the Dose Expansion Phase (Part 2) | 1 year

SECONDARY OUTCOMES:
Investigator-assessed ORR per RECIST v1.1 of IP administered AVB-001 in the Dose Escalation Phase (Part 1) | 1 year
Investigator-assessed ORR per the modified RECIST guideline for immunotherapy (iRECIST) of IP administered AVB-001 in the Dose Escalation Phase (Part 1) | 1 year
Duration of response (DOR) in the Dose Escalation Phase (Part 1) | 1 year
Progression Free Survival (PFS) in the Dose Escalation Phase (Part 1) | 1 year
Overall survival (OS) in the Dose Escalation Phase (Part 1) | 1 year
Concentrations of hIL-2 in blood and ascites/IP fluid during the Dose Escalation Phase (Part 1) | 1 year
Incidence of treatment-emergent AEs and SAEs of IP administered AVB-001 in the Dose Expansion Phase (Part 2) | 1 year
Investigator-assessed ORR per iRECIST of IP administered AVB-001 in the Dose Expansion Phase (Part 2) | 1 year
DOR in the Dose Expansion Phase (Part 2) | 1 year
PFS in the Dose Expansion Phase (Part 2) | 1 year
OS in the Dose Expansion Phase (Part 2) | 1 year
Concentrations of hIL-2 in blood and ascites/IP fluid during the Dose Expansion Phase (Part 2) | 1 year

OTHER OUTCOMES:
Immunologic changes in peripheral blood and IP environments in the Dose Escalation and Dose Expansion Phases (Parts 1 and 2) | 1 year (Part 1); 1 year (Part 2)
Analysis of anti-drug antibodies (ADA) to AVB-001 in human serum in the Dose Escalation and Dose Expansion Phases (Parts 1 and 2) | 1 year (Part 1); 1 year (Part 2)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No